CLINICAL TRIAL: NCT02849795
Title: Evaluation of Adipokines and Fat Tissue in Psoriasis and Psoriatic Arthritis and Assessment of Their Relations With the Risk of Cardiovascular Disease
Brief Title: Evaluation of Adipokines and Fat Tissue in Psoriasis and Psoriatic Arthritis
Acronym: ADIPSO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ADIPSO
Record Dates: First submitted 2016-07-27; First posted 2016-07-29 (Estimated); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Psoriasis; Arthritic Psoriasis
Keywords: Obesity, Abdominal; Adipokines; Risk of cardiovascular diseases
MeSH Terms: conditions — Psoriasis; Arthritis, Psoriatic; Obesity, Abdominal | interventions — Surveys and Questionnaires; Biological Oxygen Demand Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Psoriasis and arthritic psoriasis (Experimental): additional blood sample for biological analyses bone densitometry questionnaires
  Interventions: Other: bone densitometry; Other: questionnaires; Other: biological analyses

INTERVENTIONS:
Other: bone densitometry
Other: questionnaires
Other: biological analyses

SUMMARY:
Body composition analysis and especially body fat distribution in regions of interest (android and in particular intra-abdominal region) provides some information on the risk of cardiovascular disease. There is little data available on the body composition analysis in psoriasis and psoriatic arthritis (diseases with higher risk of cardiovascular disease), in particular data on fat distribution in regions of interest regarding the risk of cardiovascular disease.

Adipokines, secreted by the adipose tissue, have pro or anti-inflammatory and metabolic properties that are interesting to explore in pathologies with a higher risk of cardiovascular disease like psoriasis or psoriatic arthritis.

Adipokines have been investigated in psoriasis but fat tissue and in particular its distribution (android/visceral or intra-abdominal) has not been studied in parallel. Moreover, relation between adipokines and psoriasis area or severity has been studied but the relation between adipokines and cardiovascular risk factors has not yet been investigated.

The aim of this study is to investigate relations between the body fat distribution, adipokines rates and the risk of cardiovascular disease of these patients.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of psoriasis vulgaris or psoriasis pustulosa confirmed by a dermatologist or a diagnosis of psoriatic arthritis (CASPAR criteria) confirmed by a rheumatologist
* Age ≥ 18 and ≤ 80 years old
* Control group: patients matching with sex, age ± 5 years, BMI (4 groups), coming to the same hospital for a consultation.

(BMI groups : BMI < 18,5 kg/m²; 18,5 ≤ BMI ≤ 24,99 kg/m²; 25≤ BMI ≤ 29,99 kg/m²; BMI ≥ 30 kg/m²) Control group patients for psoriatic arthritis will be included during a rheumatologist consultation. They may have a non-inflammatory common disco-vertebral pathology (lumbago, lumbosciatic, spinal stenosis, neck pain, cervical arthritis and cervicobrachial neuralgia).

Control group patients for psoriasis will be included during a dermatologist consultation. They may have a non-inflammatory skin disease (acne, acne rosacea, idiopathic Raynaud's phenomenon, basal cell carcinoma, acanthosis nigricans).

In case of recruitment difficulties, healthy volunteers can be included.

* Postmenopausal women (for at least 24 months), surgically sterilized, or for women of childbearing age, efficacy use of contraceptive methods (contraceptive pills, injections or patches, intra-uterine device, double-barrier contraception),
* Signature of informed consent form
* French social security Affiliation

Exclusion Criteria:

* Pregnant woman
* Corticosteroid therapy >10 mg of prednisone or equivalent /day
* Patients taking biological therapy (anti-TNFalpha therapy: infliximab, etanercept, adalimumab, golimumab, certolizumab ; anti-Interleukin-12/Interleukin-23: ustekinumab).
* Legal incapacity or limited legal capacity
* Presence of any condition hampering compliance with the study protocol, at the discretion of the investigator
* No french social security affiliation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2014-04; Primary Completion 2017-10-17 (Actual); Study Completion 2017-10-17 (Actual)

PRIMARY OUTCOMES:
Android fat distribution measured by bone densitometry (DEXA) (LUNAR GE iDXA device) | day 1

SECONDARY OUTCOMES:
Body fat | day 1
body masses | day 1
Intra-abdominal body fat mass (measured by CoreScan) | day 1
Gynoid distribution of body fat | day 1
SCORE (Systematic COronary Risk Evaluation). | day 1
levels of adipokines | day 1
Homeostasis model assessment of insulin resistance | day 1
Bone mineral density of rachis, femoral neck, whole body | day 1
levels of ghrelin | day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Chru Besancon, Besançon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Toussirot E, Aubin F, Desmarets M, Wendling D, Auge B, Gillard J, Messica O, Guillot X, Laheurte C, Monnet E, Dumoulin G. Visceral adiposity in patients with psoriatic arthritis and psoriasis alone and its relationship with metabolic and cardiovascular risk. Rheumatology (Oxford). 2021 Jun 18;60(6):2816-2825. doi: 10.1093/rheumatology/keaa720. PMID 33232483